CLINICAL TRIAL: NCT06023472
Title: A Randomized Comparison of Microfluidic Chip vs Density Gradient Centrifugation on the Euploidy Rate of Pre-implantation Genetic Testing
Brief Title: Microfluidic Chip vs Density Gradient Centrifugation on the Euploidy Rate of Pre-implantation Genetic Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Ernest Hung-Yu Ng (Other)
Responsible Party: Sponsor-Investigator, Professor Ernest Hung-Yu Ng, Clinical Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 23-297
Record Dates: First submitted 2023-06-29; First posted 2023-09-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Infertility; Genetic Disease; Chromosomal Rearrangement; Aneuploidy
Keywords: microfluidic chip; density gradient centrifugation; euploidy rate; pre-implantation genetic testing
MeSH Terms: conditions — Infertility; Genetic Diseases, Inborn; Aneuploidy | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Intervention Model Description: On the day of oocyte retrieval, recruited women will be randomly assigned into one of the following two groups according to a computer-generated randomization list with a 1:1 ratio and a block size of 10. The randomization list will be prepared by a designated research nurse who is not involved in care of the women and opened by a laboratory staff.
  1. The microfluidic chip group and
  2. The density gradient centrifugation group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On the day of oocyte retrieval, recruited women will be randomly assigned into one of the following two groups according to a computer-generated randomization list with a 1:1 ratio and a block size of 10. The randomization list will be prepared by a designated research nurse who is not involved in care of the women and opened by a laboratory staff.
  1. The microfluidic chip group and
  2. The density gradient centrifugation group
  The women and clinicians will be blinded to the treatment groups they are assigned. Only the laboratory staff in the IVF laboratory performing sperm preparation will be aware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- The microfluidic chip group (Experimental): The Sperm Separation Device - ZyMōt Multi 850µL or 3 mL device (ZyMōt Fertility, Inc) will be used according to the volume of the raw semen samples. The microfluidics chamber will be used based on the manufacturer's instructions. 850 μL (850 μL device) or 3 mL (3mL device) of the semen sample will be added to the inlet port of the device and 750 μL (850 μL device) or 2.4 mL (3 mL device) of fertilization media will be added to the outlet port. The device will then be incubated in 6% CO2 at 37°C. After 30 minutes, 500 μL (850 μL device) or 1 mL (3mL device) of the prepared sample at the outlet port will be removed and pipetted into a labelled test tube.
  Interventions: Device: microfluidic chip
- The density gradient centrifugation group (Active Comparator): After liquefaction, sperm preparation will be completed by a discontinuous density gradient centrifugation method, using Pureception (CooperSurgical, Denmark) sperm density gradient media. The resulting sperm pellet after centrifugation will be washed once with the sperm washing medium (G-IVF Plus, Vitrolife, Sweden) The washed spermatozoa will be resuspended with the same medium, adjusting the final volume to 0.5 mL.
  Interventions: Device: density gradient centrifugation

INTERVENTIONS:
Device: microfluidic chip — Microfluidic chip method has been used for sperm sorting in order to select the most motile and morphologically normal sperm for use in assisted reproductive technologies (ART) such as in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI).
  Arms: The microfluidic chip group
Device: density gradient centrifugation — Density-gradient centrifugation is a commonly used method for sperm separation and purification. It is a technique that involves layering a semen sample on top of a gradient of different densities of a solution, typically a mixture of colloidal silica and sucrose, and then centrifuging the sample. The centrifugal force causes the sperm to migrate through the gradient, where they become separated based on their density.
  Arms: The density gradient centrifugation group

SUMMARY:
Infertile women attending for PGT at the Centre of Assisted Reproduction and Embryology, Queen Mary Hospital and Kwong Wah Hospital will be recruited during ovarian stimulation for IVF. Subsequently, they will be randomly assigned on the day of oocyte retrieval by a laboratory staff into one of the following two groups in a 1:1 ratio : (1) the microfluidic chip group and (2) the density gradient centrifugation group for sperm preparation and subsequent use in fertilization. Other IVF procedures will be the same as the standard practice of the Centre. Both women and clinicians will be blinded from the group allocation i.e. a double blind study.

DETAILED DESCRIPTION:
The study aims to investigate the treatment of couples undergoing in vitro fertilization (IVF). Eligible couples will be recruited for the study after providing informed written consent following counseling. The IVF protocol involves various steps. Women will undergo preimplantation genetic testing (PGT) as clinically indicated. Ovarian stimulation will be carried out using gonadotropin injections, and regular ultrasound monitoring will be conducted to track the growth of follicles. To prevent a premature LH surge, progestin primed ovarian stimulation or a GnRH antagonist will be administered. Once at least three follicles reach a size of over 17 mm, a trigger injection of either human chorionic gonadotrophin or a GnRH agonist will be given to induce final maturation. Oocyte retrieval will be performed 36 hours after the trigger under transvaginal ultrasound guidance.

The recruited women will be randomly assigned to one of two groups: the microfluidic chip group or the density gradient centrifugation group. Randomization and blinding will be ensured to maintain the integrity of the study. Only the laboratory staff involved in sperm preparation will be aware of the group assignment, while the women and clinicians will be blinded to the treatment groups.

Semen specimens will be collected by masturbation on the day of oocyte retrieval, following a period of 2-7 days of sexual abstinence. The semen samples will undergo evaluation according to WHO guidelines, including semen volume, sperm concentration, and percent motile spermatozoa. Sperm DNA damage will be assessed using an alkaline single-cell gel electrophoresis (Comet) assay. The extent of DNA damage in spermatozoa will be examined using specific parameters.

Sperm preparation will be performed based on the randomization list. In the microfluidic chip group, the Sperm Separation Device will be used, and the prepared sample will be collected in a test tube. In the density gradient centrifugation group, sperm preparation will be completed using a discontinuous density gradient centrifugation method, and the resulting sperm pellet will be washed and resuspended.

Oocytes will be fertilized through intracytoplasmic sperm injection, and normal fertilization will be confirmed by the presence of two pronuclei. A few cells will be taken from the blastocysts for comprehensive chromosome analysis. Cryopreservation of all blastocysts will be done, and only euploid blastocysts without aneuploidies will be replaced in subsequent frozen embryo transfer cycles.

Frozen embryo transfer (FET) will be performed in subsequent natural or hormonal replacement cycles, depending on the women's menstrual cycle regularity.

Pregnancy outcomes will be monitored through urine pregnancy tests and transvaginal ultrasounds. If the pregnancy test is positive, further ultrasounds will be done to confirm fetal viability and the number of fetuses. Pregnancy and delivery data will be retrieved after delivery, and information on pregnancy outcomes, number of babies born, birth weights, and obstetric complications will be recorded.

The study aims to assess the effectiveness of the two different sperm preparation methods and their impact on IVF outcomes, including pregnancy rates and obstetric complications.

ELIGIBILITY:
Inclusion Criteria:

* Women aged <43 years at the time of ovarian stimulation for IVF
* Women undergoing PGT for monogenic diseases, structural rearrangement of chromosomes or aneuploidy
* Sperm concentration of the raw semen with at least 0.15 million motile sperm per ml or 100 motile sperm per 50 low power field (200x) of observation

Exclusion Criteria:

* Use of frozen semen for insemination
* Use of donor oocytes and spermatozoa
* Submucosal fibroid or hydrosalpinx shown on pelvic scanning and not surgically treated;
* Women who had been recruited into this study before and
* Women joining other randomized trials

Max Age: 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 318 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Euploid rate of blastocysts | 3 months
  Euploid rate of blastocysts biopsied

SECONDARY OUTCOMES:
Live birth rate of the first embryo transfer | 3 years
  No. of live birth beyond 22 weeks of gestation per the first embryo transfer
Positive urine pregnancy test rate per the first embryo transfer | 3 years
  No. of positive urine pregnancy test per the first embryo transfer
Clinical pregnancy rate of the first embryo transfer | 3 years
  No. of clinical pregnancy per the first embryo transfer defined as presence of intrauterine gestational sac on scanning at gestational week 6.
Ongoing pregnancy rate | 3 years
  No. of ongoing pregnancy as presence of a fetal pole with pulsation at 8-10 weeks of gestation
Miscarriage rate pregnancy | 3 years
  No. of miscarriage defined as a clinically recognized pregnancy loss before the 22 weeks of pregnancy and whose denominator is the clinical pregnancy.
Multiple pregnancy rate | 3 years
  Multiple pregnancy rate: presence of more than one intrauterine sac at 6 weeks of gestation
DNA fragmentation | 3 years
  Measurement of DNA fragmentation by Comet assay using the Olive tail moment as the quantitative metric.
Ectopic pregnancy rate | 3 years
  No. of ectopic pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication of the primary paper
Access Criteria: reasonable request